CLINICAL TRIAL: NCT01185691
Title: RELIEF I: Investigating the Role of IMPELLA 2.5 System In Acutely Decompensated Chronic Heart Failure Patients. A Prospective, Single Center Feasibility Study
Brief Title: Investigating the Role of Impella 2.5 System in Acutely Decompensated Chronic Heart Failure Patients
Acronym: RELIEF I
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Low enrollment
Sponsor: Abiomed Inc. (Industry)
Collaborators: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 09-248-SDR
Record Dates: First submitted 2010-08-19; First posted 2010-08-20 (Estimated); Last update posted 2013-05-03 (Estimated); Status verified 2013-05

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Impella 2.5 — Impella 2.5 implant in patients with acute decompensated heart failure

SUMMARY:
The primary objective of this study is to assess safety and feasibility of IMPELLA 2.5 in Acute Decompensated Heart Failure patients.

ELIGIBILITY:
Major Inclusion Criteria:

1. Chronic heart failure patients, hospitalized due to decompensated heart failure (ADHF) with NYHA Class III-IV symptoms (ADHF is defined by the presence of at least one of the following symptoms/signs: dyspnea w/orthopnea, jugular venous distension, peripheral edema +2, abdominal ascites, signs of CHF on chest X-Ray)
2. LVEF ≤ 40 % within the past 3 months

Major Exclusion Criteria:

1. Acute Q-wave myocardial infarction or Acute coronary syndrome within past 30 days
2. Cardiac surgery within the past 30 days
3. Implantation of cardiac resynchronization device within past 30 days or a possibility of implanting a biventricular pacer within 90 days of randomization

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2010-07; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Major Adverse Events | 30 day or discharge(whichever is longer)

CONTACTS AND LOCATIONS:
Overall Officials: Renzo Cecere, MD, Principal Investigator — McGill University Health Centre/Research Institute of the McGill University Health Centre